CLINICAL TRIAL: NCT02796755
Title: Effects of Riluzole on CNS Glutamate and Fatigue in Breast Cancer Survivors With High Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Andrew H Miller, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00086271
Record Dates: First submitted 2016-06-02; First posted 2016-06-13 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Inflammation; Fatigue
Keywords: Central Nervous System (CNS) Glutamate; Breast Cancer Treatment; Fatigue; Cognitive Dysfunction; Behavioral; Psychometrics; Imaging Technology; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Inflammation; Fatigue; Cognitive Dysfunction; Behavior | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Riluzole Arm (Experimental): Participants will take a daily oral dose of 100 mg of riluzole (50 mg two times per day). Participants will be instructed to take the study medication on an empty stomach (1 hour before or 2 hours after meals).
  Interventions: Drug: Riluzole
- Placebo Arm (Placebo Comparator): Participants will take a daily oral dose of 100 mg of a placebo that appears identical to riluzole (50 mg two times per day). Participants will be instructed to take the study medication on an empty stomach (1 hour before or 2 hours after meals).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riluzole — Study participants randomized to this arm will take 100 mg/day of riluzole for 8 weeks.
  Other Names: Rilutek
  Arms: Riluzole Arm
Drug: Placebo — Study participants randomized to this arm will take a placebo, that matches the appearance of 100 mg tablets of riluzole, daily for 8 weeks.
  Arms: Placebo Arm

SUMMARY:
The goal of the proposed research is to determine whether riluzole, a drug that increases glutamate reuptake, will decrease central nervous system (CNS) glutamate in breast cancer survivors with increased inflammation and fatigue. The researchers will also determine whether decreasing glutamate with riluzole will reverse inflammation-related fatigue and other symptoms including cognitive dysfunction and decreased motivation. To accomplish these goals, the researchers plan to conduct an 8 week, double-blind, randomized control trial of riluzole (100 mg/d) versus placebo in 40 breast cancer survivors (n=20 per group). All breast cancer survivors will have completed treatment within 1-3 years and have a fatigue level of ≥4 (on a 10 point scale) and a plasma c-reactive protein (CRP) concentration >3mg/L (indicative of high inflammation). Participants will undergo magnetic resonance spectroscopy (MRS) to measure CNS glutamate before and after 2 and 8 weeks of riluzole or placebo treatment. Fatigue and other behavioral assessments including measures of cognitive function and motivation will be conducted before and after treatment and correlated with the change in CNS glutamate.

DETAILED DESCRIPTION:
Breast cancer is one of the most common cancers among women with ~250,000 new cases diagnosed in the US each year. Significant advances have been made in treating breast cancer, and the current number of women in the US who are considered breast cancer survivors is over 2 million. Despite these advances, breast cancer and its treatment comes at a considerable cost for a significant percentage of women with up to 30% of women experiencing behavioral and/or cognitive symptoms months to years after treatment completion. The mechanisms which contribute to these symptoms are only beginning to be understood, however, mounting data suggest that inflammation may be involved.

Prior research has demonstrated significant relationships between inflammatory markers and inflammatory signaling pathways and symptoms of fatigue and cognitive dysfunction in patients with multiple forms of cancer including breast cancer. There are a number of theories as to how inflammation may influence fatigue and cognition function in breast cancer patients. One neurotransmitter pathway that may be involved is glutamate. Inflammatory cytokines have been shown to decrease glutamate reuptake and increase glutamate release from astrocytes.

The primary objective of this study is to provide the first data on the role of CNS glutamate and symptoms of fatigue in breast cancer patients using MRS and a medication that has been shown to lower CNS glutamate in animal models and human subjects. No previous study has examined the potential connection between increased inflammation, increased CNS glutamate and symptoms in breast cancer patients, although there is strong clinical and preclinical support for an important interrelationship among these variables. Identification of a significant relationship between increased CNS glutamate and symptoms will:

* Enable the development of inflammatory biomarkers to identify patients with altered CNS glutamate.
* Help focus future studies using glutamate stabilizing medications and glutamate antagonists on patients most likely to respond to glutamate-targeted therapies (personalization of trials and treatment).
* Expand treatment studies to include synergistic or sequential targeting of inflammation and glutamate to reduce symptom burden in breast cancer patients.

This study will also serve as a foundation for efforts to link the impact of inflammatory cytokines and their relationship with increased CNS glutamate and behavior to a variety of cancers. Moreover, by testing novel treatment approaches (targeting glutamate), this study may ultimately improve the quality of life of breast cancer and other cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed surgery for Stage I-III breast cancer (lumpectomy or mastectomy) with or without neoadjuvant or adjuvant chemotherapy and with or without radiation.
* Must be 1-5 years post-treatment for breast cancer
* Must have a plasma c-reactive protein (CRP) level of >3mg/L
* Must have a score of ≥4 (out of 10 points, 0 being no fatigue and 10 being severe, incapacitating fatigue) on a Single Item Screening Scale for Fatigue

Exclusion Criteria:

* Presence of a medical condition that might represent a risk for riluzole treatment, including history of allergic reaction to riluzole and evidence of liver disease
* Presence of a medical condition that might potentially confound the relationship among CNS glutamate, inflammation and behavior/cognition, including autoimmune or inflammatory disorders, chronic infectious diseases (e.g. HIV, hepatitis B or C), pregnancy, neurologic disorders (including a history of serious head trauma or seizures), liver disease (as manifested as an elevation in liver transaminases) and uncontrolled cardiovascular, metabolic, pulmonary or renal disease (as determined by medical history and laboratory testing)
* Current or past history of schizophrenia
* Individuals with bipolar disorder who have experienced a manic episode within 6 months of study entry, or at the discretion of the study doctor
* Individuals receiving antidepressants, mood stabilizers, antipsychotic medications or benzodiazepines or drugs known to affect the immune system (e.g. glucocorticoids, methotrexate), or at the discretion of the study doctor
* Individuals exhibiting signs of infection at the screening visit will be rescheduled to screen when symptoms have resolved

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H Miller, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled beginning April 2016 and all follow-up visits were complete by October 24, 2019. Participants were enrolled from the patient population at the Emory University Winship Cancer Institute in Atlanta, Georgia.
Groups:
- Riluzole Arm: Participants took a daily oral dose of 100 mg of riluzole (50 mg two times per day) for 8 weeks. Participants were instructed to take the study medication on an empty stomach (1 hour before or 2 hours after meals).
- Placebo Arm: Participants took a daily oral dose of 100 mg of a placebo that appears identical to riluzole (50 mg two times per day), for 8 weeks. Participants will be instructed to take the study medication on an empty stomach (1 hour before or 2 hours after meals).
Period: Overall Study
Arm/Group | Riluzole Arm | Placebo Arm
Started | 15 | 15
Completed | 13 | 15
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riluzole Arm | Placebo Arm | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (6.7) | 53.7 (5.3) | 53.9 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 7 | 18
  White | 4 | 8 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Central Nervous System (CNS) Glutamate Measured by Magnetic Resonance Spectroscopy (MRS)
Description: Magnetic resonance spectroscopy (MRS) is a specialized technique associated with magnetic resonance imaging (MRI). MRS is a non-invasive way to obtain biochemical information about the tissues of the human body. Participants underwent single voxel (3-dimensional volume X pixel) MRS to measure CNS glutamate before and after 1 and 8 weeks of riluzole or placebo treatment. Voxels were placed in the right and left basal ganglia and the dorsal anterior cingulate cortex (dACC), well known targets of inflammatory cytokines on the brain, and cytokine effects on these brain regions have been associated with symptoms of fatigue and cognitive dysfunction as well as reduced motivation. MRS has shown that chronic exposure to the inflammatory cytokine interferon (IFN)-alpha leads to increased CNS glutamate (as reflected by the glutamate/creatine (Glu/Cr) ratio) which correlated with symptoms of fatigue and cognitive dysfunction.
Time Frame: Baseline, Week 1, Week 8
Measure: Mean (Standard Deviation); unit: Glu/Cr
Arm/Group | Riluzole Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
Glu/Cr
  Baseline dorsal anterior cingulate cortex (dACC) | 1.26 (0.09) | 1.2 (0.15)
  Week 1 dACC | 1.26 (1.26) | 1.27 (0.12)
  Week 8 dACC | 1.27 (0.12) | 1.27 (0.07)
  Baseline left basal ganglia | 0.85 (0.09) | 0.91 (0.12)
  Week 1 left basal ganglia | 0.93 (0.16) | 0.96 (0.13)
  Week 8 left basal ganglia | 0.96 (0.2) | 0.98 (0.11)
  Baseline right basal ganglia | 0.9 (0.09) | 0.92 (0.14)
  Week 1 right basal ganglia | 0.9 (0.08) | 0.89 (0.11)
  Week 8 right basal ganglia | 0.93 (0.13) | 0.93 (0.1)

2. Secondary Outcome: Multidimensional Fatigue Inventory (MFI) Score
Description: The Multidimensional Fatigue Inventory (MFI) is a 20-item scale used to evaluate the presence and severity of fatigue among subjects by self-reports. The MFI assesses 5 dimensions of fatigue, including general fatigue, physical fatigue, mental fatigue, reduced activity, and reduced motivation. Participants respond to fatigue related statements using a 5 point scale where 1 = "yes, that is true" and 5 = "no, that is not true". Total scores range from 20 to 100 and higher scores indicate greater fatigue.
Time Frame: Baseline, Weeks 1, 2, 4, 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riluzole Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 66.90 (10.99) | 58.90 (13.86)
  Week 1 | 63.80 (12.10) | 53.50 (15.80)
  Week 2 | 62.00 (14.60) | 53.21 (16.85)
  Week 4 | 61.07 (12.40) | 51.14 (15.64)
  Week 8 | 58.92 (16.47) | 46.50 (13.85)

3. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Fatigue Short Form Score
Description: PROMIS-Fatigue Short Form is a 7-item scale developed by the Patient-Reported Outcome Measurement Information System (PROMIS), a part of the NIH Roadmap Initiative which is focused on developing a publicly available resource of standardized, accurate, and efficient outcome measures of symptoms, distress, and functioning. The criterion for a minimally clinically important difference in patients with advanced-stage cancer is a 3 to 5 point difference in raw score. Recommendations for high priority research on cancer-related fatigue recommend use of the PROMIS fatigue scale to allow comparison of results across studies. Respondents indicate how much they agree with the item statements on a scale from 1 (not at all) to 5 (very much). Total scores range from 7 to 35 with higher scores indicating greater fatigue.
Time Frame: Baseline, Weeks 1, 2, 4, 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riluzole Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 25.1 (3.8) | 21.8 (5.0)
  Week 1 | 22.5 (4.3) | 18.71 (5.06)
  Week 2 | 23.7 (5.5) | 17.07 (6.18)
  Week 4 | 21.6 (5.8) | 17.36 (6.07)
  Week 8 | 18.8 (6.1) | 15.07 (6.11)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time consent to participate in the study was given through the Week 8 study visit.
Arm/Group | Riluzole Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 11/15 | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riluzole Arm (N=15) | Placebo Arm (N=15)
Headache (General disorders) | 4 (4) | 2 (2)
Gastrointestinal distress (Gastrointestinal disorders) | 6 (6) | 3 (3)
Itch/Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 1 (1)
Paresthesia (General disorders) | 0 (0) | 1 (1)
Increased white blood cell count (General disorders) | 0 (0) | 1 (1)
Venipuncture complications (Surgical and medical procedures) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT02796755/Prot_SAP_000.pdf